CLINICAL TRIAL: NCT05475600
Title: Adapted Physical Activity and Relaxation by Biofeedback in Patients With Haematological Malignancy Admitted in Intensive Care unit_APAER_H Protocol
Brief Title: APA and Relaxation by Biofeedback in Patients With Haematological Malignancy Admitted in ICU
Acronym: APAER_H
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-01-CHRMT
Record Dates: First submitted 2022-07-13; First posted 2022-07-27 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Adapted Physical Activity; Hematological Malignancies; Anxiety; Relaxation
MeSH Terms: conditions — Hematologic Neoplasms; Anxiety Disorders | interventions — Glutamyl Aminopeptidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Classical APA group (Experimental): Activity type: aerobic Frequency: 3 sessions per week Duration of session: 30 to 60 min Intensity: mild to moderate (4-6 on Rated Perceived Exertion (RPE) Scale) Session description: 1 - Warm-up 5 to 10 min / Activation of devices and systems: muscular, articular, cardiovascular / Objective: preparation of body and mind for physical activity. 2 - Training 10 to 30 min physical activity with à classical cyclo-ergometer 3 - Cool down 15 to 20 min / stretching / Objective: to bring the body back to a resting state
  Interventions: Behavioral: Classical APA group:
- APA with Exergaming device (Experimental): Activity type: aerobic Frequency: 3 sessions per week Duration of session: 30 to 60 min Intensity: mild to moderate (4-6 on RPE Scale) Session description: 1 - Warm-up 5 to 10 min / Activation of devices and systems: muscular, articular, cardiovascular / Objective: preparation of body and mind for physical activity. 2 - Training 10 to 30 min physical activity with à classical cyclo-ergometer 3 - Cool down 15 to 20 min / stretching / Objective: to bring the body back to a resting state
  Interventions: Behavioral: APA with Exergaming device
- APA associated with biofeedback relaxation (Experimental): Activity type: aerobic Frequency: 3 sessions per week Duration of session: 30 to 60 min Intensity: mild to moderate (4-6 on RPE Scale) Session description: 1 - Warm-up 5 to 10 min / Activation of devices and systems: muscular, articular, cardiovascular / Objective: preparation of body and mind for physical activity. 2 - Training 10 to 30 min physical activity with an Exergaming device 3 - Cool down: 20 min / Biofeedback relaxation device / Objective: to bring the body back to a resting state
  Interventions: Behavioral: APA associated with biofeedback relaxation

INTERVENTIONS:
Behavioral: Classical APA group: — Activity type: aerobic Frequency: 3sessions per week Duration of session: 30 to 60min Intensity: mild to moderate (4-6 on RPE Scale) Session description: 1 - Warm-up 5 to 10min / Activation of devices and systems: muscular, articular, cardiovascular / Objective: preparation of body and mind for physical activity. 2 - Training 10 to 30min physical activity with à classical cyclo-ergometer 3 - Cool down 15 to 20min / stretching / Objective: to bring the body back to a resting state
  Arms: Classical APA group
Behavioral: APA with Exergaming device — Activity type: aerobic Frequency: 3sessions per week Duration of session: 30 to 60min Intensity: mild to moderate (4-6 on RPE Scale) Session description: 1 - Warm-up 5 to 10min / Activation of devices and systems: muscular, articular, cardiovascular / Objective: preparation of body and mind for physical activity. 2 - Training 10 to 30min physical activity with à classical cyclo-ergometer 3 - Cool down 15 to 20min / stretching / Objective: to bring the body back to a resting state
  Arms: APA with Exergaming device
Behavioral: APA associated with biofeedback relaxation — Activity type: aerobic Frequency: 3sessions per week Duration of session: 30 to 60min Intensity: mild to moderate (4-6 on RPE Scale) Session description: 1 - Warm-up 5 to 10min / Activation of devices and systems: muscular, articular, cardiovascular / Objective: preparation of body and mind for physical activity. 2 - Training 10 to 30min physical activity with à Exergaming device 3 - Cool down: 20min / Biofeedback relaxation device / Objective: to bring the body back to a resting state
  Arms: APA associated with biofeedback relaxation

SUMMARY:
Adapted Physical Activity (APA) is accepted as an effective, recommended and beneficial supportive care for the health of people with cancer during the different phases of the disease. The objective of the project is to analyse the effect of APA programs (Classic, Exergaming and Relaxation) on the state anxiety of people with severe blood diseases admitted to Intensive Care Unit (ICU). Anxiety is a major affect in this context. The interest of the practice of APA for this public is to reduce the level of state anxiety and to limit the decline of functional capacities. The main objective of this work is to identify whether specific and/or complementary effects result from the use of biofeedback and/or Exergaming.

DETAILED DESCRIPTION:
Haematological malignancies have several unpleasant consequences on psychological and physical health. Indeed, an important fatigue and reduction of functional capacities appear. Reduction of functional capacities leads to the reduction of autonomy in Acts of Daily Living (ADL) and impact negatively the global Quality of Life (GQoL). Patients who undergo high dose treatment in protected area have higher risks of functional decline. In addition, hospital stay alone in sterile room favours increase of anxiety and depression.

Health care strategies are going to integrate and use more of support care as APA and relaxation. Regular APA practice leads to maintain and/or improve physical functioning and psychological well-being. Physical Activity ensures to maintain or develop muscular strength and cardio-respiratory capacities that patients loose if they stay inactive during hospital stay. APA practice participates too in regulation of emotional states. Indeed, it favours positive emotions as self-esteem, self-confidence, satisfaction and pleasure. In the order to limit or reduce anxiety level, relaxation provides an effective response. Maintain functional capacities and reduce negatives emotional states participate to reduce fatigue too. Also, APA associated with relaxation seems to be a good effective support care strategy.

The aim of this study is to implement a supervised APA program with entertaining devices as Exergaming and Biofeedback relaxation for patients undergo high dose treatment in protected area.

Exergaming consists on exercise and training through fun or recreative situations.

Biofeedback device is a relaxation tool that gives feedback on functioning of nervous system in real time. The objective is to leads patients to become aware of their body-information to finally, associate them to sensations and more effectively control them.

The objectives of this study are to:

1. To reduce state anxiety level and psychological fatigue impact on GQoL and
2. To Maintain or improve functional capacities and reduce physical fatigue.

The main hypotheses are:

1. Each of the three programs leads to the objectives specified above.
2. APA associated with biofeedback relaxation reduce more state anxiety level than APA with Exergaming that is more effective than APA classic.
3. APA with Exergaming and biofeedback practice gender more satisfaction and adhesion than APA classic

The program takes place 3 times per week. Each session lasts between 30 and 60 min. Intensity of effort is defined as light to moderate. Participants are assigned to one of the tree groups: 1-APA classic / 2-APA with Exergaming / 3-APA and Biofeedback relaxation. Aerobic activity is performed on a cyclo-ergometer (Groups 1 and 3) classic or exergaming (group 2). At the end of session, patients in relaxation group (Group 3) realise relaxation as recovery whereas other groups rest and stretch.

Functional capacities are assessed twice by submaximal tests: at the beginning and directly after APA program, just before hospital discharge. The first session affords to estimate subjects capacities and to create and individualised and adapted programme. The second affords to compare groups themselves and each other. Cardio-respiratory capacity is evaluated by the 2min Walk Test (2WT) and lower limbs muscular strength by the 5 Times Sit to Stand Test (FTSST). State anxiety level and fatigue are assessed by State and Trait Anxiety Inventory-YA (STAI-YA) and Multi-Fatigue Inventory_20items (MFI-20) respectively. At the inclusion, we complete the profile of individuals with the Hospital Anxiety and Depression Scale (HADS).

Adhesion and satisfaction are assessed by feedbacks of participants and by the comparison of the number of planned versus performed sessions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 75 years old
* Admitted in Intensive Care Unit
* Informed consent

Exclusion Criteria:

* Contraindication for physical exercise
* Inability to understand the French language (written and/or oral)
* Ongoing involvement in another proprietary research protocol
* Lack of affiliation to social security

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in State Anxiety by the State Trait Anxiety Inventory - YA Version | 2 moments: at the beginning and directly at the end of program.
  Self-reported questionnaire with 20 items assessed on a 4 points scale

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | Once at the inclusion
  14 items Questionnaire to detect anxiety and depressive disorders
2min Walk Test (2MWT) | : twice: at the beginning of the study and at the end: immediately after the APA program
  sub-maximal test to assess functional capacity
Sit to Stand Test (SST) | twice: at the beginning of the study and at the end: immediately after the APA program
  Sub-maximal test to assess muscular strength
Multi-Fatigue Inventory_20 items (MFI-20) | Twice: at the beginning of the study and at the end: just before hospital discharge.
  20-item scale designed to evaluate five dimensions of fatigue: general fatigue, physical fatigue, reduced motivation, reduced activity, and mental fatigue.
EORTC quality of life questionnaire quality of life questionnaire (QLQ)-C30 | Twice: At the beginning of the study and one month after the intervention
  Questionnaire developed to assess the quality of life of cancer patients
Evaluation of the acute effect of an adapted physical activity session on the change in state Anxiety by the State Trait Anxiety Inventory - YA Version | Twice at each moment: just before the session and directly after it to obtain the acute effect of the APA Session.
  Self-reported questionnaire with 20 items assessed on a 4 points scale

OTHER OUTCOMES:
Analysis of blood balance data | twice: at the beginning of the study and at the end: immediately after the APA program.
  Immune system activity by using the results of blood samples performed as part of the usual care protocol.
  Data analysed include:
  * Polynuclear neutrophils rate
  * Leukocyte rate
  * Hemoglobin rate
  * Platelets rate
  * Haematocrit rate

CONTACTS AND LOCATIONS:
Overall Officials: Véronique DORVAUX, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France

REFERENCES:
- [Derived] Bousmia J, Langlet C, Elnar AA, Goetz C, Bolmont B, Dorvaux V. Adapted physical activity, exergaming and relaxation by biofeedback in haematological intensive care unit in France: study protocol of a randomised controlled trial (APAER-H trial). BMJ Open. 2025 Dec 4;15(12):e099876. doi: 10.1136/bmjopen-2025-099876. PMID 41344711